CLINICAL TRIAL: NCT05504629
Title: Characterizing The Interindividual Postexercise Hypotension Response For Two Order of Concurrent Training In Patients With Morbid Obesity
Brief Title: Interindividual Postexercise Hypotension Response in Morbid Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional Andres Bello (Other)
Collaborators: Universidad de La Frontera (Other)
Responsible Party: Principal Investigator, Cristian Alvarez, Principal investigator, Universidad Nacional Andres Bello
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UNAB-FCR-KINE2022A
Record Dates: First submitted 2022-08-13; First posted 2022-08-17 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Metabolic Syndrome; Morbid Obesity
MeSH Terms: conditions — Metabolic Syndrome; Obesity, Morbid | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endurance Training (ET) plus Resistance Training (RT) (Experimental): Concurrent training of Endurance Training plus Resistance Training order.
  Interventions: Behavioral: RT+ET
- Resistance Training (RT) plus Endurance Training (ET) (Active Comparator): Concurrent training of Resistance Training plus Endurance Training order.
  Interventions: Behavioral: Concurrent training order 1

INTERVENTIONS:
Behavioral: Concurrent training order 1 — atag
  Other Names: Exercise training
  Arms: Resistance Training (RT) plus Endurance Training (ET)
Behavioral: RT+ET — aetaer
  Other Names: Concurrent training order 2
  Arms: Endurance Training (ET) plus Resistance Training (RT)

SUMMARY:
A quasi-experimental study developed in sedentary morbidly obese men and women (age 43.6±11.3 y; body mass index [BMI] ≥40 kg/m2) were assigned to a CT group of ET plus RT (ET+RT; n=19; BMI 47.8±16.7) or RT plus ET order group (RT+ET; n=17; BMI 43.0±8.0). Subjects of both groups received eight exercise sessions over four weeks. Systolic (SBP), diastolic (DBP), mean arterial pressure [MAP], heart rate at rest [HR], and pulse pressure [PP] measurements before and after 10 minutes postexercise. Secondary outcomes were other anthropometric, body composition, metabolic, and physical condition parameters. Using the ∆SBP reduction, and quartile categorization (Q) in 'high' (Rs: quartile 4), 'moderate' (MRs: quartile 3), 'low' (LRs: quartile 2), and 'nonresponders' (NRs: quartile 1) were reported.

DETAILED DESCRIPTION:
Independent of the order (i.e., ET+RT, or RT+ET), each CT session had two sections; RT and ET, which were applied two days per week, during 8 sessions (4 weeks), and where the blood pressure changes were measured only in four opportunities (i.e., once a week in sessions 2, 4, 6, and 8). Thus, the CT included in each session 3 stages; a) callisthenics exercises, b) main exercise (ET+RT or RT+ET), and c) cool down exercises.

Before the starting, the participants were involved in the maximum strength capacity estimated using a submaximal test based on the Brzycki's equation: weight [1.0278-(0.0278*repetitions)] that does not change based on the sex, age of the population, or the exercise modality that is performed (Mayhew et al., 2004). After this procedure, there were applied 4 familiarization sessions that consisted in; session 1: 'knowledge of all measurements', 'knowledge of exercise-machine manipulation', and 'instructions during the exercise program', session 2: 'exercising during cycling', 'weights, and metal bars', session 3: 'applying a few of exercises of RT in 2 to 3 sets of exercises, to know the configuration of each exercise (i.e., ET and RT regimes itself), and session 4: 'applying the 50 to 70% of their CT program' corresponding to a normal session compound. In the 'calisthenic stage', each subject developed 10 minute warm-up with continuous walking, joint mobility and flexibility exercises. In the 'main part' of the session, and independent of the CT order group (ET+RT or RT+ET), the ET section consisted of continuous cycling using a magnetic resistance static bicycle (OxfordTM Fitness, model BE-2701, Chile) for 20 minutes. The intensity of the ET exercise was regulated through the previously used modified Borg scale from 1 to 10 rating of perceived exertion (Gillen et al., 2013) and the participants worked at a level between 5 to 7 points (i.e., moderate-intensity), considering the original 6 to 20 points scale (Borg, 1998), being the subjects regularly controlled to not exceed this intensity restriction. On the other hand, the RT section included 8 to 12 muscle strength exercises of circuit training with the following different muscle groups: (1) forearm, (2) knee flexors and extensors, (3) trunk, (4) chest, (5) shoulder elevators, (6) horizontal shoulder flexors, (7) extensors, and finally (8) plantar flexors. These exercises were performed in one set in a continuous concentric/eccentric voluntary contraction as possible for 60 seconds, followed by 60 to 90 seconds of passive recovery, where each participant was changed to another exercise. The RT section was of 25 minutes in duration time.

ELIGIBILITY:
Inclusion Criteria:

* age >18 and <60 years
* women or men
* medical authorization for physical tests
* body mass index (BMI) ≥40 kg/m2, or between 35 and 40 kg/m2 but with previously diagnosed of morbid obesity and candidate for bariatric surgery

Exclusion Criteria:

* physical limitations to performing the physical test (e.g., restrictive injuries of the musculoskeletal system)
* exercise-related dyspnoea or respiratory alterations
* chronic heart disease diagnosed during the time of morbid obesity diagnosed and the starting of the exercise intervention

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2019-10-05 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure measured by a blood pressure cuff | From baseline to 10 minutes after exercise training
  Change from Baseline in systolic blood pressure in the unit of (mmHg)
Diastolic blood pressure measured by a blood pressure cuff | From baseline to 10 minutes after exercise training
  Change from Baseline in diastolic blood pressure in the unit of (mmHg)
Mean arterial pressure measured by a blood pressure cuff | From baseline to 10 minutes after exercise training
  Change from Baseline in mean arterial blood pressure in the unit of (mmHg)

SECONDARY OUTCOMES:
Heart rate at rest measured by a cardiometer watch | From baseline to 10 minutes after exercise training
  Change from Baseline in Heart rate at rest in (beats per minute)
Pulse pressure measured by a blood pressure cuff | From baseline to 10 minutes after exercise training
  Change from Baseline in Pulse pressure in the unit of (mmHg)
Body mass measured by a scale | From baseline to 10 minutes after exercise training
  Change from Baseline in Body mass in (kg)
Body mass index calculated from weight plus height and elevated to square | From baseline to 10 minutes after exercise training
  Change from Baseline in Body mass index in (kg/m2)
Waist circumference measured by a flexible tape | From baseline to 10 minutes after exercise training
  Change from Baseline in Waist circumference in (cm)
Body fat percentage measured by a digital bioimpedanciometer scale | From baseline to 10 minutes after exercise training
  Change from Baseline in Body fat percentage in (%)
Lean mass measured by a digital bioimpedanciometer scale | From baseline to 10 minutes after exercise training
  Change from Baseline in Body fat percentage in (kg)
Skeletal muscle mass measured by a digital bioimpedanciometer scale | From baseline to 10 minutes after exercise training
  Change from Baseline in Skeletal muscle mass in (kg)
Bone mass measured by a digital bioimpedanciometer scale | From baseline to 10 minutes after exercise training
  Change from Baseline in Bone mass in (kg)
Basal metabolic rate measured by a digital bioimpedanciometer scale | From baseline to 10 minutes after exercise training
  Change from Baseline in Basal metabolic rate in (Kcal)
Fasting plasma glucose measured by blood sample in fasting state | From baseline to 10 minutes after exercise training
  Change from Baseline in Fasting plasma glucose in (mg/dL)
Total cholesterol measured by blood sample in fasting state | From baseline to 10 minutes after exercise training
  Change from Baseline in Total cholesterol in (mg/dL)
Low density lipids measured by blood sample in fasting state | From baseline to 10 minutes after exercise training
  Change from Baseline in Low density lipids in (mg/dL)
High density lipids measured by blood sample in fasting state | From baseline to 10 minutes after exercise training
  Change from Baseline in High density lipids in (mg/dL)
Triglycerides measured by blood sample in fasting state | From baseline to 10 minutes after exercise training
  Change from Baseline in Triglycerides in (mg/dL)
Six minutes walking test measured by a walking test into a sport court | From baseline to 10 minutes after exercise training
  Change from Baseline in Six minutes walking test in (m)
Handgrip muscle strength of the non-dominant arm measured by a dynamometer hand equipment | From baseline to 10 minutes after exercise training
  Change from Baseline in Handgrip strength in the non-dominant arm measured by dynamometer at sitting position in (kg)
Handgrip strength Dominant arm measured by a dynamometer hand equipment | From baseline to 10 minutes after exercise training
  Change from Baseline in Handgrip strength in the Dominant arm measured by dynamometer at sitting position in (kg)

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Delgado Floody, PhD, Principal Investigator — Universidad de La Frontera
Locations (1):
- Universidad de La Frontera, Temuco, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Delgado-Floody P, Izquierdo M, Ramirez-Velez R, Caamano-Navarrete F, Moris R, Jerez-Mayorga D, Andrade DC, Alvarez C. Effect of High-Intensity Interval Training on Body Composition, Cardiorespiratory Fitness, Blood Pressure, and Substrate Utilization During Exercise Among Prehypertensive and Hypertensive Patients With Excessive Adiposity. Front Physiol. 2020 Oct 19;11:558910. doi: 10.3389/fphys.2020.558910. eCollection 2020. PMID 33192554
- [Result] Delgado-Floody P, Soriano-Maldonado A, Rodriguez-Perez MA, Latorre-Roman PA, Martinez-Salazar C, Vargas CA, Caamano-Navarrete F, Jerez-Mayorga D, Alvarez C. The Effects of Two Different Concurrent Training Configurations on Markers of Metabolic Syndrome and Fitness in Women With Severe/Morbid Obesity: A Randomised Controlled Trial. Front Physiol. 2021 Sep 21;12:694798. doi: 10.3389/fphys.2021.694798. eCollection 2021. PMID 34621181
- [Result] Alvarez C, Ramirez-Campillo R, Ramirez-Velez R, Izquierdo M. Effects and prevalence of nonresponders after 12 weeks of high-intensity interval or resistance training in women with insulin resistance: a randomized trial. J Appl Physiol (1985). 2017 Apr 1;122(4):985-996. doi: 10.1152/japplphysiol.01037.2016. Epub 2017 Feb 2. PMID 28153946

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-17): https://cdn.clinicaltrials.gov/large-docs/29/NCT05504629/Prot_SAP_001.pdf